CLINICAL TRIAL: NCT00776022
Title: An Open Label, Randomized, Single-center, Single-dose, Two-treatment, Two-period, Crossover Bioavailability Study Comparing Cetirizine Hydrochloride 10 mg Tablet of Ohm Laboratories Inc. (A Subsidiary of Ranbaxy, Inc) With Zyrtec® Cetirizine Hydrochloride, 10 mg Tablet of Pfizer Labs (Division of Pfizer Inc.) in Healthy, Adult, Human Subjects Under Fed Condition
Brief Title: Bioequivalence Study of Cetirizine Hydrochloride 10mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Collaborators: Ohm Laboratories, Inc. (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Laboratories Limited
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 11849
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Healthy
Keywords: Bioequivalence Cetirizine Hydrochloride 10 mg tablet fed conditions
MeSH Terms: interventions — Cetirizine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cetirizine Hydrochloride 10 mg tablet of Ohm Laboratories
  Interventions: Drug: Cetirizine Hydrochloride 10 mg tablet
- 2 (Active Comparator): Cetirizine Hydrochloride 10 mg tablet of Pfizer Labs
  Interventions: Drug: Cetirizine Hydrochloride 10 mg tablet

INTERVENTIONS:
Drug: Cetirizine Hydrochloride 10 mg tablet — Bioequivalence Cetirizine Hydrochloride 10 mg tablet fed conditions

SUMMARY:
An open label, randomized, single-center, single-dose, two-treatment, two-period, crossover bioavailability study comparing Cetirizine Hydrochloride 10 mg tablet of Ohm Laboratories Inc. (A subsidiary of Ranbaxy, Inc) with Zyrtec® Cetirizine Hydrochloride, 10 mg tablet of Pfizer Labs (Division of Pfizer Inc.) in healthy, adult, human subjects under fed condition

DETAILED DESCRIPTION:
The study was conducted as an open label, randomized, single-center, single-dose, two-treatment, two-period, crossover bioavailability of the test formulation of cetirizine hydrochloride tablet of Ohm Laboratories Inc. (A subsidiary of Ranbaxy, Inc) containing 10 mg cetirizine hydrochloride study comparing to the marketed product, Zyrtec®, containing 10 mg of cetirizine hydrochloride of Pfizer Labs (Division of Pfizer Inc.), in healthy, adult, human, subjects under fed condition.

Safety measures were performed throughout the study and included a physical examination, laboratory evaluation, and measurement of vital signs.

A total of 32 subjects were randomized to receive single oral dose of cetirizine hydrochloride 10 mg tablet and 29 subjects completed both the periods of the study.

ELIGIBILITY:
Inclusion Criteria:

* - Aged 18-50 years.
* Were within 18 to 29.9 kilograms/m2 per the BMI (Determination of Body Mass Index).
* Had voluntarily given written informed consent to participate in this study.
* Were of normal health as determined by medical history and physical examination of the subjects performed within 30 days prior to the commencement of the study.
* Blood chemistry, hematology, and urinalysis tests performed within 30 days prior to the start of the study must be within clinically acceptable limits upon evaluation by the Investigator.
* Subjects must have screening and check-in (each period) blood pressure and pulse rate within the protocol specified ranges.
* If female and of childbearing potential, the subject was counseled on the importance of not becoming pregnant before or during the study, and the subject had a negative pregnancy test at the pre-treatment visit.

Exclusion Criteria:

* - History of clinically significant organ-system (cardiovascular, neurological, hepatic, hematopoietic, pulmonary, endocrine, or gastrointestinal) disorders, or ongoing infectious diseases.
* history of alcohol abuse or drug addiction requiring treatment within the last 12 months.
* Presence or history of renal impairment or chronic liver disease.
* History of jaundice (yellowing of the skin or whites of the eyes).
* Participation in an investigationaldrug study or donation of blood within 30 days prior to the start of the study.
* Known allergy or sensitivity to cetirizine (Zyrtec®), or to related drugs such as hydroxyzine (Vistaril® or Ataraxl®).
* Prescription drug use (excluding hormonal contraceptives) within 14 days prior to drug administration, each period. Subject is taking macrolide antibiotics, such as erythromycin, azithromicin, ketoconazole, or related drugs.
* Ingestion of grapefruit juice or grapefruit-containg products within 72 hours prio to drug administration, each period.
* Alcohol consumption 24 hours prior to drug administration, each period.
* Caffeine or xanthine consumption for at least 10 hours prior to drug administration, each period.
* Female subjects who are pregnant or nursing.
* Positive HIV 1, Hepatitis B surface antigen, and urine screen for drugs of abuse within 30 days prior to the start of the study.

Ages: 18 Years to 50 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2005-04; Primary Completion 2005-04 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of Bioequivalence between ranbaxy acetaminophen 650 mg extended release gelcaps and Tylenol® Arthritis Pain extended release caplets (containing acetaminophen 650 mg) of Mc Neil-PPC Inc.,under fed conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Bioanalytical Systems, Inc, Baltimore, Maryland, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html